CLINICAL TRIAL: NCT04548089
Title: Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) - Empowering Resilience and Holistic Wellbeing for Sustaining Family Caregiving: A Waitlist Randomized Controlled Trial
Brief Title: Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) : A Waitlist Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Principal Investigator, Nanyang Technological University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-2019-05-021
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Caregiver Burnout; Caregiver Stress
Keywords: Dementia Caregiving, Caregiver Stress, Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Upon referrals made by the collaborating institutions and other community dementia-care organizations, consenting caregivers will be allocated to either the immediate treatment group or wait-list control group. Baseline assessment [T1] is conducted through face-to-face interviews, or self-administered questionnaires, facilitated by the research team.
  Participants assigned to the treatment group will then attend a 4-week MCAT-DC programme conducted jointly by an experienced mindfulness practitioner and a credentialed art therapist or artist. Thereafter, immediate post intervention assessment [T2] will be carried out, with follow-up assessments at 4 weeks [T3], 3-months [T4] and 6-month [T5]. Participants assigned to the wait-list control group will be assessed at second baseline [T2], thereafter, attend a 4-week MCAT-DC programme, followed by an immediate post intervention assessment [T3], as well as follow-up assessments at 3-months [T4] and 6-months [T5].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants assigned to the immediate intervention group will engage in a 4-week 2.5-hour Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) with intervention elements of brief psycho-education, weekly mindfulness meditation, facilitated creative art making, reflective writing, group sharing and discussion.
  Interventions: Behavioral: Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC)
- Waitlist Control Group (Experimental): Participants assigned to the wait-list control group will not receive Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) until one month after baseline assessment.
  Interventions: Behavioral: Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC)

INTERVENTIONS:
Behavioral: Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) — Each Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) will focus on 3 major areas that cultivate self-care, resilience and communal support. The specific intervention structure include: Week 1 - Empowering Self-Care: Introduction to the science of stress, self-care, burnout, as well as the arts and mindfulness to cultivate resilience; Week 2 - Reflective Caregiving: Reflection of caregiving experiences that demonstrates strengths and challenges; Week 3 - Understanding Loss: Introduction to the science of loss, how grief can impair hope and wellbeing, and how self-compassion can help transform suffering into blessings.; Week 4 - Meaning Reconstruction: Reflection on caregiver identities, to elicit the lessons and wisdoms learnt, and to create renewed meaning to sustain their caregiving journeys. Guided mindfulness mediation will also be professionally recorded to form a daily take-home mindfulness mediation exercise for participants, each exercise will last 10-20 minutes.

SUMMARY:
The current study builds on the empirical foundation of Mindful-Compassion Art Therapy (MCAT) to test its efficacy as a multicomponent, holistic, psycho-socio-spiritual intervention for supporting dementia family caregivers. MCAT is a group-based intervention that integrates mindfulness meditation and art therapy, with reflective awareness complementing emotional expression, to foster self-compassion and inner-resilience among professional caregivers. A wait-list RCT design is adopted to refine and extend the application of MCAT to empower self-care and resilience among 102 dementia family caregivers recruited via community-based dementia-care organizations in Singapore. The expected outcomes will advance theory and practice for sustainable dementia family caregiving in Singapore and around the globe.

DETAILED DESCRIPTION:
Background: Dementia is a neurodegenerative disease that leads to irreversible decline in one's cognitive and functional capacity, identity, and personhood. In Singapore, the number of persons with dementia is expected to soar to 187,000 by 2050. Hence, it is imperative to render comprehensive support to dementia sufferers, and especially their family caregivers. While local initiatives have raised public awareness and developed services for dementia care, they do not adequately address the psycho-socio-spiritual needs of family caregivers, as caregiving stress can greatly impede one's mental and emotional health. International research for dementia family caregivers has thus focused on developing multicomponent interventions that accentuate holistic support to promote healthy and sustainable caregiving.

Objective and Methods: Building on the established MCAT protocol (Ho et al., 2019), this study will adopt a wait-list randomized controlled trial design to test the efficacy of the refined version of Mindful-Compassion Art Therapy for Dementia Care (MCAT-DC) among 102 dementia family caregivers in Singapore. This study aims to: 1) develop a disease-specific version of MCAT for Dementia Care (MCAT-DC); 2) assess MCAT-DC's effectiveness in reducing caregiver stress and burden; 3) assess MCAT-DC's effectiveness for reducing caregivers' depressive symptoms and psychophysiological distress, while enhancing resilience, hope, spirituality, meaning and quality-of-life; and 4) assess the feasibility and acceptability of a standardized MCAT-DC protocol for large-scale implementation.

Significance: MCAT is an effective psycho-social-spiritual intervention for reducing stress and promoting holistic wellbeing among professional caregivers. It has received wide recognition and distinction among palliative care and research communities for its clinical innovation and effectiveness. Given the robust evidence on MCAT's positive impact on professional caregivers, it is anticipated that a refined version of MCAT will have similar, if not greater, benefits for family caregivers. The study findings will form new knowledge to advance both theory and practice for sustainable dementia family caregiving in Singapore and around the globe.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver of a family member with diagnosed with dementia
* Fluent in written and verbal english

Exclusion Criteria:

* Unable to provide informed consent
* Diagnosed with major mental conditions or cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in scores on Caregiver Distress (HADS) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Caregiver Distress is assessed using the Hospital Anxiety and Depression Scale (HADS), a 14-item scale that evaluates levels of anxiety and depression (Zigmond & Snaith, 1983; Snaith, 2003)
Change in scores on Caregiver Burden (ZBI-12) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Caregiver burden is assessed by the Zarit Burden Interview-Short (ZBI-12), a 12-item self-reported questionnaire comprising of three subscales of role-strain, self-criticism, and negative emotions (Tang et al., 2016).

SECONDARY OUTCOMES:
Change in scores on Depressive Symptoms (PHQ-4) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Depressive symptoms is assessed by the Patient Health Questionnaire (PHQ-4), a reliable and widely used self-reported scale (Kroenke, 2009).
Change in scores on Resilience (ER89-R) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Trait resilience is assessed by the 10-item Ego-Resilience Revised Scale (ER-89R) (Alessandri et al., 2011).
Change in scores on Hope (HHI) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Hope is assessed by the 12-item Herth Hope Index (HHI) (Herth, 1992).
Change in scores on Spirituality (FACIT-Sp) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Spirituality is assessed by the Peace and Meaning sub-scales (8-items) of the 'Functional Assessment of Chronic Illness Therapy - Spiritual Wellbeing Scale' (FACIT-Sp) (Bredle et al., 2011).
Change in scores on Support with Grief (ISS) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Perceived social support with grief is measured with a modified version of the 5-item 'Inventory of Social Support' (ISS). This scale assesses an individual's satisfaction with their social support networks (Hogan & Smidt, 2002).
Change in scores on Quality of Life (WHOQoL-8) from baseline | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  The 8-item World Health Organization Quality of Life Scale-8 (WHOQoL-8) is used to assess subjective quality of life (da Rocha et al., 2012).

OTHER OUTCOMES:
Heart Rate Variability | Baseline [T1], Immediately after completion of the intervention/control protocol [T2], One month post intervention/control protocol [T3], Three months post intervention/control protocol [T4], six months post intervention/control protocol [T5].
  Heart Rate Variability (HRV), a reliable biomarker that reflects an individual's cardiovascular stress regulation, is used to assess participants' psychophysiological well-being (Wheat & Larkin, 2010). Ithlete, a small non-invasive portable HRV measurement device, together with a smart tablet installed with the ithlete HRV App, is used for this assessment. Concisely, an Infrared Pulse Plethysmography finger sensor is attached to participants' index finger while following a series of brief breathing instruction on the screen of the smart tablet, and during this 1-2 minute exercises, data of their psychophysiological performance are collected.

CONTACTS AND LOCATIONS:
Overall Officials: Andy HY Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (3):
- Singapore (3):
  - Tan Tock Seng Hospital (Centre for Geriatric Medicine), Singapore
  - Tan Tock Seng Hospital (Department of Palliative Medicine), Singapore
  - Khoo Teck Puat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alessandri G, Vecchione M, Caprara G, Letzring TD. The ego resiliency scale revised. European Journal of Psychological Assessment. 2011 Nov 28.
- [Background] da Rocha NS, Power MJ, Bushnell DM, Fleck MP. The EUROHIS-QOL 8-item index: comparative psychometric properties to its parent WHOQOL-BREF. Value Health. 2012 May;15(3):449-57. doi: 10.1016/j.jval.2011.11.035. Epub 2012 Feb 9. PMID 22583455
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Ho AHY, Tan-Ho G, Ngo TA, Ong G, Chong PH, Dignadice D, Potash J. A novel mindful-compassion art therapy (MCAT) for reducing burnout and promoting resilience for end-of-life care professionals: a waitlist RCT protocol. Trials. 2019 Jul 8;20(1):406. doi: 10.1186/s13063-019-3533-y. PMID 31287010
- [Background] Hogan NS, Schmidt LA. Testing the grief to personal growth model using structural equation modeling. Death Stud. 2002 Oct;26(8):615-34. doi: 10.1080/07481180290088338. PMID 12243195
- [Background] Bredle JM, Salsman JM, Debb SM, Arnold BJ, Cella D. Spiritual well-being as a component of health-related quality of life: the functional assessment of chronic illness therapy-spiritual well-being scale (FACIT-Sp). Religions. 2011 Mar;2(1):77-94.
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Tang JY, Ho AH, Luo H, Wong GH, Lau BH, Lum TY, Cheung KS. Validating a Cantonese short version of the Zarit Burden Interview (CZBI-Short) for dementia caregivers. Aging Ment Health. 2016 Sep;20(9):996-1001. doi: 10.1080/13607863.2015.1047323. Epub 2015 May 27. PMID 26016419
- [Background] Wheat AL, Larkin KT. Biofeedback of heart rate variability and related physiology: a critical review. Appl Psychophysiol Biofeedback. 2010 Sep;35(3):229-42. doi: 10.1007/s10484-010-9133-y. PMID 20443135
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Ho AHY, Tan-Ho G, Ngo TA, Ong G, Chong PH, Dignadice D, Potash J. A Novel Mindful-Compassion Art-Based Therapy for Reducing Burnout and Promoting Resilience Among Healthcare Workers: Findings From a Waitlist Randomized Control Trial. Front Psychol. 2021 Oct 21;12:744443. doi: 10.3389/fpsyg.2021.744443. eCollection 2021. PMID 34744918